CLINICAL TRIAL: NCT06777745
Title: Improvement of Breast Examination Skills of Midwifery Students: Model Supported Education Study
Brief Title: Model Supported Breast Examination Training for Midwifery Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Merve AKINCI, Assistant Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-77192459-050.99-376938; KBÜBAP-24-ABP-160 (Other: Scientific Research Projects)
Record Dates: First submitted 2024-12-20; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Breast Self-Examination; Midwifery Students Education; Clinical Competence; Self-Confidence
Keywords: Midwife; student; breast examination; model
MeSH Terms: conditions — Breast Self-Examination

STUDY DESIGN:
Who Masked: Participant
Masking Description: The students were not informed about the groups they were in. Single blind was provided in the study by knowing which group they would be in by the researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Model-assisted breast examination application (Experimental): After obtaining consent from the students in the experimental group, pre-test data will be collected by filling out the 'Personal Information Form,' 'Self-Confidence Scale,' and 'Student Satisfaction and Confidence in Learning Scale. After the theoretical information is given, the examination stages will be shown practically on the breast examination model in the laboratory environment. Students taken in groups of 10 will be examined and evaluated one by one after the lecture; 15 minutes will be allocated to each student. Two weeks later, the students will reapply all the examination steps in the laboratory, and the missing steps will be identified and completed by the researcher. In this process, 'Self-Confidence Scale' and 'Student Satisfaction and Confidence in Learning Scale' will be completed for the post-test. Two weeks later, the same scales will be applied again for the final post-test.
  Interventions: Other: Model-assisted breast examination application
- Control group (No Intervention): After obtaining consent from the control group students, pre-test data will be collected using the 'Personal Information Form,' 'Self-Confidence Scale,' and 'Student Satisfaction and Confidence in Learning Scale.' Students will then receive theoretical instruction and watch a video detailing examination stages, including identifying the area, manual examination, examination methods, nipple evaluation, and detecting malignant formations. Two weeks later, students will practice the steps in a laboratory setting based on the theoretical course. During the examination, the researcher will use the 'Breast Examination Skill Assessment Form' to note complete and incomplete steps, explain missing steps, and have students complete them. The 'Self-Confidence Scale' and 'Student Satisfaction and Confidence in Learning Scale' will be re-administered as a post-test. Two weeks later, the same scales will be used for a final post-test.

INTERVENTIONS:
Other: Model-assisted breast examination application — Designed for the development of self-examination skills, this model is in the shape of a female upper body with medium-sized breasts. Thanks to its ergonomic design, it can be worn easily and offers a comfortable use. Made of high quality, dermatologically tested and tactile silicone material. This model, which reflects all the details of the skin realistically, has a structure suitable for standing and lying examination. For educational use, there are 2 benign tumours, 4 malignant tumours and 2 typical anomalies. This model allows for practical explanation of all stages of breast examination such as determining the area to be examined, manual examination of the area, examination method, nipple examination and detection of malignant formations in the breast.
  Arms: Model-assisted breast examination application

SUMMARY:
Breast cancer is the most common cancer among women worldwide and early detection significantly improves treatment success. Screening methods used for early detection include breast self-examination (BSE), clinical breast examination (CBE) and mammography. It is critical for midwifery students to learn CCM and teach this method to women. CPM allows women to recognise early signs through breast self-examination. This method is simple and inexpensive and can be applied without requiring much time and labour. Practical training of midwifery students helps them to ensure the effectiveness and correct application of this method. The use of breast examination models during the training process gives students practical experience in detecting signs of breast cancer, such as nipple depression, discharge, asymmetry of the breasts and the appearance of orange peel. In addition, midwifery students can develop their clinical skills by having the opportunity to make mistakes and gain hands-on experience in a safe environment. This process can contribute to increasing early diagnosis rates and improving treatment processes.The sample of this pre-test, post-test, follow-up randomised controlled study consisted of 64 midwifery students (experimental=32, and control=32). Data will be collected with Personal Information Form (PIF), Breast Examination Skills Assessment Form (BESAF), Self-Confidence Scale (SC) and Student Satisfaction and Confidence in Learning Scale (SCSLS). After obtaining the consent of the students in the experimental group, pre-test data will be obtained by filling out the 'Personal Information Form', 'Self-Confidence Scale' and 'Student Satisfaction and Confidence in Learning Scale'. Then, theoretical information will be given and the examination stages such as determining the area to be examined, manual examination of the area, examination method, nipple examination and detection of malignant formations in the breast will be explained practically in the breast examination model in the laboratory environment. Students will be taken in groups of 10, and after the application is explained, each student will perform the breast examination and evaluation individually. Approximately 15 minutes will be allocated for each student. Two weeks after the breast model application, the same students will be taken to the laboratory and asked to perform all the examination steps again. While the students are performing the examination steps, the researcher will mark the complete and incomplete applications on the 'Breast Examination Skill Evaluation Form' and the missing steps will be explained to the students and they will be asked to complete them. At the same time, 'Self-confidence Scale' and 'Student Satisfaction and Confidence in Learning Scale' will be filled out for the post-test. Then, two weeks later, the 'Self-Confidence Scale' and 'Student Satisfaction and Confidence in Learning Scale' will be filled out again for the final post-test. After obtaining the consent of the students in the control group, pre-test data will be collected by applying 'Personal Information Form', 'Self-Confidence Scale' and 'Student Satisfaction and Confidence in Learning Scale' to the students. Then, the students will be given theoretical information and a video will be shown to them, which includes examination stages such as determining the area to be examined, manual examination of the area, examination method, nipple examination and detection of malignant formations in the breast.

Two weeks later, the students will be taken to the laboratory environment and will be asked to perform the application steps in line with the theoretical course they have taken. While the students are performing the examination steps, the researcher will mark the complete and incomplete applications on the 'Breast Examination Skill Evaluation Form', then the missing steps will be explained to the students and they will be asked to complete them. In the post-test phase, the 'Self-Confidence Scale' and the 'Student Satisfaction and Confidence in Learning Scale' will be administered to the students again. Two weeks after this process, the same scales will be filled in again for the final post-test.

DETAILED DESCRIPTION:
Early diagnosis of breast cancer, one of the most common cancers worldwide, significantly enhances the success of treatment. It is crucial for midwifery students to learn breast self-examination and teach this technique to women. This study introduces an innovative approach to address the lack of practical experience among midwifery students. Breast examination mock-ups offer students the opportunity to practice in a safe and controlled environment, enabling them to apply their theoretical knowledge in practice. This contributes to enhancing students' clinical skills and improving their effectiveness in patient care. Moreover, the study aims to improve the quality of midwifery education by providing an effective solution to the challenges posed by limited resources and the increasing number of midwifery students.

By offering students the chance to practice in a secure environment, this study is expected to help midwifery students develop their skills and cope with the lack of clinical experience. The study aims to assess the use of breast examination models as a solution to this practical experience gap, providing students with an opportunity to refine their skills and enhance their clinical competence. The sample of this pre-test, post-test, follow-up randomised controlled study consisted of 64 midwifery students (experimental=32, and control=32). Data will be collected with Personal Information Form (PIF), Breast Examination Skills Assessment Form (BESAF), Self-Confidence Scale (SC) and Student Satisfaction and Confidence in Learning Scale (SCSLS). After obtaining the consent of the students in the experimental group, pre-test data will be obtained by filling out the 'Personal Information Form', 'Self-Confidence Scale' and 'Student Satisfaction and Confidence in Learning Scale'. Then, theoretical information will be given and the examination stages such as determining the area to be examined, manual examination of the area, examination method, nipple examination and detection of malignant formations in the breast will be explained practically in the breast examination model in the laboratory environment. Students will be taken in groups of 10, and after the application is explained, each student will perform the breast examination and evaluation individually. Approximately 15 minutes will be allocated for each student. Two weeks after the breast model application, the same students will be taken to the laboratory and asked to perform all the examination steps again. While the students are performing the examination steps, the researcher will mark the complete and incomplete applications on the 'Breast Examination Skill Evaluation Form' and the missing steps will be explained to the students and they will be asked to complete them. At the same time, 'Self-confidence Scale' and 'Student Satisfaction and Confidence in Learning Scale' will be filled out for the post-test. Then, two weeks later, the 'Self-Confidence Scale' and 'Student Satisfaction and Confidence in Learning Scale' will be filled out again for the final post-test. After obtaining the consent of the students in the control group, pre-test data will be collected by applying 'Personal Information Form', 'Self-Confidence Scale' and 'Student Satisfaction and Confidence in Learning Scale' to the students. Then, the students will be given theoretical information and a video will be shown to them, which includes examination stages such as determining the area to be examined, manual examination of the area, examination method, nipple examination and detection of malignant formations in the breast.

Two weeks later, the students will be taken to the laboratory environment and will be asked to perform the application steps in line with the theoretical course they have taken. While the students are performing the examination steps, the researcher will mark the complete and incomplete applications on the 'Breast Examination Skill Evaluation Form', then the missing steps will be explained to the students and they will be asked to complete them. In the post-test phase, the 'Self-Confidence Scale' and the 'Student Satisfaction and Confidence in Learning Scale' will be administered to the students again. Two weeks after this process, the same scales will be filled in again for the final post-test.

This study presents an innovative approach to supporting midwifery students in developing their clinical skills. The use of breast examination models enables students to better prepare for real clinical situations by applying theoretical knowledge. It is anticipated that students in the experimental group will exhibit higher levels of self-confidence and skill development compared to the control group. These findings could provide valuable data to promote the widespread adoption of model-assisted education in clinical training programs. Given the increasing number of students and the limitations of clinical facilities, model-assisted education emerges as a sustainable and effective solution to enhance the quality of midwifery programs. This method allows students to develop their skills without compromising patient safety and offers flexibility in the educational process. The study's results are expected to guide the structuring of educational programs in midwifery and other healthcare fields.

ELIGIBILITY:
Inclusion Criteria:

* Being a 2nd, 3rd or 4th year midwifery student at Karabük University Faculty of Health Sciences
* Being between the ages of 18-25
* Voluntarily agreeing to participate in the study
* Being a citizen of the Republic of Turkey

Exclusion Criteria:

* Leave whenever you want without working.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Self-confidence Scale | 2 mounth
  Self-Confidence Scale is a 33-item Likert-type scale developed by Akın (2007) to assess the self-confidence level of individuals. The scale consists of two sub-dimensions: internal self-confidence and external self-confidence. The items are scored between 1 (Never) and 5 (Always). The total score ranges from 33 to 165, with higher scores indicating higher self-confidence. Self-confidence level is evaluated by dividing the total score by the number of items: Below 2.5 is considered low self-confidence, between 2.5-3.5 is considered medium self-confidence and above 3.5 is considered high self-confidence.
Student Satisfaction and Confidence in Learning Scale | 2 mounth
  The 'Student Satisfaction and Confidence in Learning Scale' developed to measure students' attitudes and beliefs about simulation was published by the National League for Nurses. The internal consistency coefficient of the scale, whose Turkish validity and reliability was performed by Karaçay and Kaya in 2017, was found to be 0.88. The scale has two sub-dimensions as 'satisfaction with learning' and 'self-confidence' and the total number of items is 13. The scale is answered in a five-point Likert scale. The minimum score obtained from the scale is 17 and the maximum score is 61.
Breast Examination Skill Assessment Form | 3 mounth
  The form prepared by the researchers to evaluate the participants' breast self-examination skills comprehensively includes the steps, techniques and points to be considered during breast examination. The form includes questions to evaluate the basic stages of breast examination such as observation, palpation (palpation), symmetry control, nipple examination, detection of masses or suspicious formations. In this way, the level of correct and complete application of the participants during breast examination is evaluated.
Personal Information Form | 2 mounth
  The form containing questions about the socio-demographic data of the participants was prepared by the researchers.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No